CLINICAL TRIAL: NCT06218693
Title: VIA Family - Family Based Early Intervention Versus Treatment as Usual- 4 Year Follow-up
Brief Title: VIA Family 4 Year Follow-up of a Family-based Preventive Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); Child and Adolescent Mental Health Services, Research Unit, Capital Region, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHSCRDenmark_VIAFAMILY
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Mental Disorder
Keywords: Familial high-risk children; preventive psychiatry; offspring
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIA Family intervention (Experimental): VIA Family is a family based intervention. A multidisciplinary team of specialists from adult mental health services, child and adolescent mental health services and social services will be responsible for providing the basic treatment elements that are: case management and regular contact with the case manager, psychoeducation for the whole family, parental training (Triple P) and early intervention for mental problems of the child.
  Interventions: Behavioral: VIA Family
- Treatment as Usual (TAU) (Active Comparator): TAU is defined as any kind of help and support focusing on high risk children and parental mental illness within the catchment area of the study. At present, the municipalities and the mental health services do not offer any kind of family focused intervention addressing parental mental illness that can be compared to the VIA Family program.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: VIA Family — A family-based, multi-component, individual-tailored intervention based on case-management.
  Arms: VIA Family intervention
Behavioral: Treatment As Usual (TAU) — care as usual
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study aims to investigate the long-term effects (2.5 years after post-intervention) of a preventive family-based intervention (VIA Family) compared with treatment as usual (TAU) for children of parents with a severe mental illness.

Background:

Children of parents with a mental illness have an increased lifetime risk of developing a mental illness themselves. Preventive interventions for families with children with high familial risk can potentially disrupt the transgenerational transmission.

The current study is a follow-up study of a trial investigating the effect of the preventive intervention: the VIA Family trial.

The VIA Family trial investigated the superiority of a preventive family-based intervention, VIA Family, compared with treatment as usual (TAU) in improving children's, parents' and families' functioning and well-being. Eligible families had at least one parent with a lifetime severe mental illness diagnosis ( i.e. recurrent major or moderate depression, bipolar disorder, or schizophrenia spectrum disorder), at least one child between the ages of 6-12 years and lived within the Frederiksberg or Copenhagen (Denmark). The trial had a randomized, two-armed, parallel and controlled design. The participating families were randomly assigned to both groups with an allocation ratio of 1:1.

The current study is a follow-up study aiming to explore the effect of the intervention 2.5 years after post-intervention.

The main research questions for the current follow-up study are:

1. Do children participating in the VIA Family intervention experience a greater decrease in symptoms of mental illness from baseline (timepoint 0) to long-term follow-up (timepoint 2) compared with children allocated to TAU?
2. Do parents participating in the VIA Family intervention experience a greater decrease in perceived parental stress from baseline (timepoint 0) to long-term follow-up (timepoint 2) compared with parents allocated to TAU?

ELIGIBILITY:
Inclusion Criteria:

* Child must have address registered in the municipality of Frederiksberg or Copenhagen.
* At least one of the biological parents must have a diagnosis of schizophrenia spectrum disorder, bipolar affective disorder or recurrent major depression.
* The parent with a diagnosis must have had at least one in- or outpatient contact with the mental health system within the lifetime of the child.

Exclusion Criteria:

* Parents who do not speak and understand enough Danish to be able to give informed consent for their own and for the child's participation.
* If all family members are currently engaged in an intensive family intervention program addressing parental functioning and child development, they are excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in "Strength and Difficulties Questionnaire" (SDQ) | Change from baseline to 4 years follow-up
  Parent reported 25-items questionaire of their child's behavioural and emotional difficulties, 3-point Likert scale (0,1,2), higher scores indicate more emotional or behavioral problems

SECONDARY OUTCOMES:
Change in Children's Global Assessment Scale (CGAS) | Change from baseline to 4 years follow-up
  A clinician rated measurment to asses general functioning in children (scale from 1-100. High score represent better outcome)
Change in Family Assessment Device (FAD) | Change from baseline to 4 years follow-up
  A 60 item parent report questionaire assesing family functioning ( scale 1-4. Low score represent better outcome) [Time Frame: Change from baseline at 18 month follow-up]
Change in Home Observation for Measurement of the Environment (HOME) | Change from baseline to 4 years follow-up
  A clinican rated semi structured interview measuring stimulation and support in the home ( scale 0-60. High score represent better outcome)
Health-Related Quality of Life Questionnaire: KIDSCREEN -10 | Change from baseline to 4 years follow-up
  A child-rated questionnaire on Healthrelated Quality of Life., 5-point Likert Scale, score range 10-50 ( higher score better quality of life)
This is Me (TIM) | Change from baseline to 4 years follow-up
  A child-rated questionnaire on self-esteem,higher scores indicate better self-esteem
Parental Stress Scale (PSS) | Change from baseline to 4 years follow-up
  A parent-rated questionnaire on the quality of experienced stress related to parenting, score 1-5, higher score more perceived parental stress
Personal and Social Performance Scale (PSP) | Change from baseline to 4 years follow-up
  A clinician rated measurement to asses global functioning in parents, higher score indicates higher functioning
Parenting Scale (PS) | Change from baseline to 4 years follow-up
  A parent-rated questionnaire on parenting (30items) Higher scores indicate dysfunctional parenting

CONTACTS AND LOCATIONS:
Overall Officials: Anne A E Thorup, Principal Investigator — Research Unit at Child and Adolescent Mental Health Center, Capital Region, Denmark
Locations (1):
- Research Unit at Child and Adolescent Mental Health Center, Capital Region, Denmark, Hellerup, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT06218693/SAP_000.pdf